CLINICAL TRIAL: NCT05658809
Title: Total Thyroidectomy Versus Hemithyroidectomy for Patients With Single Thyroid Nodule , Prospective Comparative Study
Brief Title: Intervention in Single Thyroid Nodule.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Anter Ali Abdelhamid, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THYSINGLE
Record Dates: First submitted 2022-11-23; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Thyroidectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total thyroidectomy for single thyroid nodule (Active Comparator): group of participants will be treated with total thyroidectomy
  Interventions: Procedure: thyroidectomy
- Hemithyroidectomy for single thyroid nodule (Active Comparator): 2nd group of participants will be treated with hemithyroidectomy
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — Patients will be divided into 2 groups group will be treated with total thyroidectomy and the other group will be treated with hemithyroidectomy

SUMMARY:
Thyroid nodules are common clinical problem. The incidence is 2-4 per 100,000 people per year, being more common in women and the elderly. thyroid nodule is a "discrete lesion within the thyroid gland that is radiologically distinct from the surrounding thyroid parenchyma. Most thyroid nodules are asymptomatic, may present as neck swelling

DETAILED DESCRIPTION:
Thyroid nodular disease comprises of a wide range of disorders. Benign forms such as colloid nodules,cysts and thyroiditis are more comman than benign follicular neoplasms and thyroid carcinomas. Incidence of malignancy ranges from 10% to 30% in solitary thyroid nodule(STN).Studies have shown that the occurrence of malignancy is higher in case of solitary thyroid nodule compared to multinodular goitres. Preoperative evaluation of thyroid nodules is important in distinguishing between benign and malignant thyroid nodules and also in treatment to avoid unnecessary extensive surgery and its complications. Fine needle aspiration biopsy (FNAB) is the most common method of examining solitary thyroid nodules today.Total thyroidectomy and lobectomy remain the main primary surgical interventions for single thyroid nodule. There is debat between total thyroidectomy and hemithyroidectomy for patients with single thyroid nodule. our study is for comparing between total thyroidectomy and hemi thyroidectomy in single thyroid nodule

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 60 years.
2. patients with single thyroid lesion
3. Fit for surgery

Exclusion Criteria:

1. patients with age less than 20 years and more than 60 years.
2. patients with multiple thyroid lesions.
3. patients with advanced and metastatic malignancy.
4. Unfit for surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in the management of single thyroid nodule to reduce the morbidity and mortality rates | one year
  Compare between total thyroidectomy and hemithyroidectomy in patients with single thyroid nodule to improve the management of single thyroid nodule in general surgery department , Assiut university hospital.

REFERENCES:
- [Background] Hurtado-Lopez LM, Arellano-Montano S, Torres-Acosta EM, Zaldivar-Ramirez FR, Duarte-Torres RM, Alonso-De-Ruiz P, Martinez-Duncker I, Martinez-Duncker C. Combined use of fine-needle aspiration biopsy, MIBI scans and frozen section biopsy offers the best diagnostic accuracy in the assessment of the hypofunctioning solitary thyroid nodule. Eur J Nucl Med Mol Imaging. 2004 Sep;31(9):1273-9. doi: 10.1007/s00259-004-1544-7. Epub 2004 May 6. PMID 15133637
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Jena A, Patnayak R, Prakash J, Sachan A, Suresh V, Lakshmi AY. Malignancy in solitary thyroid nodule: A clinicoradiopathological evaluation. Indian J Endocrinol Metab. 2015 Jul-Aug;19(4):498-503. doi: 10.4103/2230-8210.159056. PMID 26180765
- [Background] Lloyd RV, Buehler D, Khanafshar E. Papillary thyroid carcinoma variants. Head Neck Pathol. 2011 Mar;5(1):51-6. doi: 10.1007/s12105-010-0236-9. Epub 2011 Jan 8. PMID 21221869
- [Background] Alwithenani R, DeBrabandere S, Rachinsky I, MacNeil SD, Badreddine M, Van Uum S. Performance of the American Thyroid Association Risk Classification in a Single Center Cohort of Pediatric Patients with Differentiated Thyroid Cancer: A Retrospective Study. J Thyroid Res. 2019 Jun 2;2019:5390316. doi: 10.1155/2019/5390316. eCollection 2019. PMID 31275541
- [Background] Popoveniuc G, Jonklaas J. Thyroid nodules. Med Clin North Am. 2012 Mar;96(2):329-49. doi: 10.1016/j.mcna.2012.02.002. PMID 22443979